CLINICAL TRIAL: NCT05203861
Title: Reward and Threat Sensitivity as Mediators of Positive and Negative Affect Treatment
Brief Title: Affect Treatment for Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Michelle Craske, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R33MH115138 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Affect Treatment (Experimental): 15 sessions of psychotherapy designed to augment reward anticipation, reward attainment, and reward learning.
  Interventions: Behavioral: Positive Affect Treatment
- Negative Affect Treatment (Active Comparator): 15 sessions of psychotherapy designed to decrease threat avoidance, threat appraisal and arousal.
  Interventions: Behavioral: Negative Affect Treatment

INTERVENTIONS:
Behavioral: Positive Affect Treatment — Sessions 1-7: Pleasurable activities + imaginal recounting and reinforcement of positive mood effects (continued for sessions 8-15) Sessions 8-10: Cognitive exercises focusing on identifying positive aspects of experience, taking responsibility for positive outcomes, and imagining future positive events Sessions 11-14: Exercises to cultivate and savor positive experiences Session 15: Relapse prevention.
  Arms: Positive Affect Treatment
Behavioral: Negative Affect Treatment — Sessions 1-7: Exposure therapy to feared or avoided situations, sensations, or memories (continued for sessions 8-15) Sessions 8-10: Cognitive restructuring of probability, cost, and attributional biases Sessions 11-14: Capnometry-assisted respiratory training Session 15: Relapse prevention
  Arms: Negative Affect Treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy and mediators of change in Positive Affect Treatment, a psychotherapy specifically aimed at enhancing reward sensitivity in individuals with low positive affect (a core feature of anhedonia) in the context of depression or anxiety.

Target enrollment is 100 male and female participants with low positive affect and depression or anxiety and impaired functioning, between the ages of 18 and 65 years, who will be randomized to either Positive Affect Treatment or Negative Affect Treatment (designed to reduce threat sensitivity). Participants will complete laboratory tests, psychiatric assessments, and self-report questionnaires as part of the study.

The total length of participation is around 5 months.

DETAILED DESCRIPTION:
Low positive affect in the context of depression or anxiety has been relatively resistant to pharmacological and psychological treatments. Newer treatments that focus upon positivity or reward sensitivity have shown promising results.

As a replication and extension of a prior NIMH funded R61 phase trial, the purpose of this R33 phase randomized controlled trial is to evaluate the efficacy and mediators of change of Positive Affect Treatment (designed to augment reward sensitivity) for individuals with low positive affect in the context of depression or anxiety symptoms. Mediators (targets) include behavioral, cognitive, physiological and experiential measures of two reward targets: reward anticipation and response to reward attainment. Specificity of target engagement is assessed by comparison with Negative Affect Treatment, designed to reduce threat sensitivity, and by including behavioral, cognitive, physiological and experiential mediators (targets) that assess threat sensitivity.

Clinical outcomes are assessed at baseline and either weekly or at Week 5, Week 10, Week 16 (post), and one-month follow-up. Mediators (targets) are assessed at baseline, Week 5, Week 10, Week 16 (post) and one-month follow-up. Mediational models will evaluate the degree to which change in the target measures explain change in the outcome measures.

Target enrollment is 100 male and female participants with low positive affect and depression or anxiety and impaired functioning between the ages of 18 and 65 who will be randomized to Positive Affect Treatment or Negative Affect Treatment, each comprising 15 individual psychotherapy sessions.

Participants will complete laboratory tests and psychiatric assessments and self-report questionnaires as part of the study. Total length of participation is around 5 months.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Low positive affect indexed by less than or equal to 24 on the positive affect subscale of the PANAS (i.e., PANAS-P); and scores of greater than or equal to 11 for depression, greater to or equal to 6 for anxiety, or greater to or equal to 10 for stress on the Depression, Anxiety, and Stress Scale; and scores of greater than or equal to 5 on any Sheehan Disability Scale subscale.
* Willingness to refrain from starting other psychosocial or pharmacological treatments until study completion.

Exclusion Criteria:

* Patient report of serious medical conditions - such as history of serious, uncontrolled medical illness, or instability (including significant cardio-pulmonary disease, organic brain syndrome, seizure disorder, cerebrovascular disease, thyroid dysfunction, and diabetes)
* Active suicidal ideation
* Lifetime history of bipolar disorder, psychosis, cognitive impairment, or organic brain damage
* Substance abuse in the last 6 months or dependence within last 12 months.
* Greater than 11 cigarettes per week or nicotine equivalent
* History of marijuana, cocaine or stimulant use 5-7 times/week or more before age 15 (e.g., amphetamine, cocaine, methamphetamine)
* Willingness to refrain from marijuana use 1 week before laboratory assessments
* Pregnancy
* Bupropion, dopaminergic or neuroleptic medications use in the past 6 months
* Heterocyclics and SSRIs are permitted if stabilized (3 months) and PRN benzodiazepines and beta-blockers are permitted but discouraged on laboratory assessment visits
* Refusal of video/audio-taping
* Prior participation in previous waves of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule Expanded (PANAS-X) (General Dimensions Scales) | Baseline to post-treatment (16 weeks) and follow-up (20 weeks)
  Reported positive affect (general dimensions scale positive affect) and negative affect (general dimension scale negative affect) (score range for each scale: 10-50, higher scores represent higher levels of positive affect or negative affect).
Depression Anxiety and Stress Scale (DASS-21) | Baseline to post-treatment (16 weeks) and follow-up (20 weeks)
  Reported symptoms of depression (score range: 0-21), anxiety (score range: 0-21), and stress (score range: 0-21), higher scores indicate higher severity and frequency.

SECONDARY OUTCOMES:
Interviewer Anhedonia Ratings | Baseline, post-treatment (16 weeks) and follow-up (20 weeks)
  Interviewer ratings of interest, pleasure, and motivation in hobbies/pastimes, foods/drinks, social activities (score range: 1-12), higher scores indicate lower anhedonia
Sheehan Disability Scale (SDS) | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Reported impairment due to symptoms (score range: 0-30) with higher scores indicating greater impairment. Includes reported number of days of missed school/work and number of days of reduced productivity.
Beck Scale for Suicide Ideation | Baseline, post-treatment (16 weeks) and follow-up (20 weeks)
  Reported suicidal ideation (score range: 0-38), higher scores indicate higher suicidality
Positive and Negative Affect Schedule Expanded (PANAS-X) Basic Positive Emotions Scales and Serenity | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: Reported positive affect (basic positive emotions scales and serenity) (score range: 19 - 95). Note: items which overlap with the general dimensions scale for positive affect (see Outcome 1) will not be included in this composite score. Excluded overlapping items include: alert, attentive, determined, enthusiastic, excited, proud, and strong.
Effort-Expenditure for Rewards Task (EEfRT) | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: behavioral effort for reward
Monetary Incentive Task | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: cardiac acceleration to anticipation of reward
Behavioral Inhibition/Behavioral Activation (reward drive subscale) (BAS-RD) | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: Reported reward sensitivity (score range: 4-16), and threat sensitivity (score range: 7-28), with higher scores indicating higher sensitivity
Dimensional Anhedonia Rating Scale | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: Reported reward desire, motivation, effort, and pleasure (score range: 0-68), with higher scores indicating higher degree of reward desire, motivation, effort, and pleasure
Modified Attentional Dot Probe Task | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: attentional engagement with positive and negative stimuli
International Affective Picture System Task | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: cardiac response to positive stimuli
Temporal Experience of Pleasure Scale (consummatory subscale) | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: Reported reward consummatory pleasure (score range: 8-48)
Anxiety Sensitivity Index | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: Reported threat appraisal of anxiety (score range: 0-64)
Probability and Cost Questionnaire for Social and Physical Outcomes | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: Reported threat appraisal of social and physical outcomes (score range: 0-80 for each subscale), with higher scores indicating higher cost/probability estimation
Mental Arithmetic Task | Baseline, Week 5, Week 10, post-treatment (Week 16) and follow-up (Week 20)
  Mediator: cardiorespiratory response to stress

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Southern Methodist University, Dallas, Texas

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT05203861/Prot_SAP_ICF_000.pdf